CLINICAL TRIAL: NCT05127746
Title: An Open-label, Randomized, Cross-over, Multiple Dose, Phase 1 Clinical Trial to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of DA-5207 Transdermal Delivery System in Healthy Adults
Brief Title: Phase 1 Clinical Trial of DA-5207 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA5207_AD2_Ib
Record Dates: First submitted 2021-11-05; First posted 2021-11-19 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Healthy
MeSH Terms: interventions — Donepezil; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Period 1, Aricept 5mg → DA-5207 A; Period 2, Aricept 5mg → Aricept 10mg
  Interventions: Drug: Aricept 5mg Tablet; Drug: Aricept 10mg Tablet; Drug: DA-5207 A
- Sequence 2 (Experimental): Period 1, Aricept 5mg → Aricept 10mg; Period 2, Aricept 5mg → DA-5207 A
  Interventions: Drug: Aricept 5mg Tablet; Drug: Aricept 10mg Tablet; Drug: DA-5207 A
- Sequence 3 (Experimental): Period 1, Aricept 5mg → DA-5207 B; Period 2, Aricept 5mg → Aricept 10mg
  Interventions: Drug: Aricept 5mg Tablet; Drug: Aricept 10mg Tablet; Drug: DA-5207 B
- Sequence 4 (Experimental): Period 1, Aricept 5mg → Aricept 10mg; Period 2, Aricept 5mg → DA-5207 B
  Interventions: Drug: Aricept 5mg Tablet; Drug: Aricept 10mg Tablet; Drug: DA-5207 B

INTERVENTIONS:
Drug: Aricept 5mg Tablet — 1 tablet once daily
Drug: Aricept 10mg Tablet — 1 tablet once daily
Drug: DA-5207 A — 1 patch once weekly
  Arms: Sequence 1; Sequence 2
Drug: DA-5207 B — 1 patch once weekly
  Arms: Sequence 3; Sequence 4

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics and pharmacodynamics of DA-5207 transdermal delivery system in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Health Volunteers (Age: 19~55 years)
* Body Weight: Male≥55kg, Female≥50kg
* 18.5 ≤BMI≤ 25.0

Exclusion Criteria:

* Galactose intolerance, Lapp lactase deficiency, Glucose-galactose malabsorption
* Allergy or Drug hypersensitivity
* Clinically significant Medical History
* AST, ALT>Upper Normal Range*1.25, eGFR<60mL/min/1.73m²
* Heavy caffeine intake
* Heavy alcohol intake (more than 210g/week)
* Heavy smoker (more than 10 cigarettes/day)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
AUC | 29-36 days
  area under the concentration-time curve
Css,max | 0-36 days
  maximum serum concentration at steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Jeonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea